CLINICAL TRIAL: NCT00904137
Title: Taping Versus Splinting Versus Above Elbow Casting for Type I Supracondylar Fractures of the Humerus in Children: A Randomized Controlled Trial
Brief Title: Treatment of Type I Supracondylar Fractures of the Humerus
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We were unable to recruit the appropriate numbers as parents did not want to randomize their child for the treatments options.
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Kishore Mulpuri, Principle Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H08-02904
Record Dates: First submitted 2009-05-15; First posted 2009-05-19 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Type I Supracondylar Fracture of the Humerus
Keywords: Supracondylar fracture; humerus; elbow
MeSH Terms: interventions — POLR1G protein, human; Splints

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cast (Active Comparator): Above elbow fiberglass cast with a collar-and-cuff
  Interventions: Procedure: Cast
- Splint (Active Comparator): Long arm posterior plaster splint with a collar-and-cuff
  Interventions: Procedure: Splint
- Tape (Active Comparator): Elastoplast tape applied to keep the elbow in flexion, with a collar-and-cuff
  Interventions: Procedure: Tape

INTERVENTIONS:
Procedure: Cast
  Arms: Cast
Procedure: Splint
  Arms: Splint
Procedure: Tape
  Arms: Tape

SUMMARY:
Type I supracondylar fractures are elbow fractures that occur in children aged 3-10 years. Many different treatment options exist to treat this type of fracture. The purpose of this study is to compare three different treatment modalities with regards to pain experienced during treatment, the amount of pain medication needed during treatment, and any short-term complications. We hypothesize that above elbow casting and long-arm splinting will result in less pain and have fewer complications than taping the elbow in flexion.

DETAILED DESCRIPTION:
Patients who meet the inclusion criteria will be enrolled into the study either by the attending physician in the Emergency Department at BC Children's hospital or by one of the study investigators. They will be randomly assigned to one of three treatment groups: above elbow cast, long arm splint, or tape. After being treated, patients will be required to fill in a daily pain diary describing their level of pain and how much analgesia they are requiring. They will also be followed by regular phone calls to track any complications of treatment (e.g. loosening or shifting of cast/ splint/ tape, any skin breakdown, etc.). Patients will be seen for follow-up at three weeks post-injury in the Orthopedics Clinic at BCCH to have radiographs repeated, finish their treatment, and hand in their pain diaries.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 4-12 years who present to the Emergency department at BC Children's hospital with a history of elbow trauma, and are diagnosed by the staff emergency physician to have a Type I supracondylar fracture of the humerus (as seen on AP and lateral radiographs of the elbow)

Exclusion Criteria:

* patients with neurovascular compromise associated with the fracture
* a pre-existing diagnosis of metabolic or structural bone disease that predisposes them to fractures
* presence of other fractures of the ipsilateral upper extremity

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2009-05; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Mean pain intensity and median pain duration over treatment period | 3 weeks

SECONDARY OUTCOMES:
Amount of analgesia required during treatment period, incidence of complications associated with treatment | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kishore Mulpuri, Principal Investigator — University of British Columbia; Renjit Varghese, Study Director — University of British Columbia; Lisa Dyke, Study Director — University of British Columbia; Firoz Miyanji, Study Director — University of British Columbia; Christopher Reilly, Study Director — University of British Columbia
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada